CLINICAL TRIAL: NCT03870347
Title: Prospective Evaluation of Opiate Use Status in Patients Referred for Endoscopic Evaluation of Bile Duct Dilation
Brief Title: Opiate Use and Biliary Dilation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Subhas Banerjee, Associate Professor of Medicine, Stanford University
Other Study IDs: 45243
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Evaluation of Association Between Opiate Use and Biliary Dilation
MeSH Terms: interventions — Endosonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Biliary Dilation Cohort: Patients referred for endoscopic evaluation of biliary dilation
  Interventions: Diagnostic Test: Endoscopic ultrasound

INTERVENTIONS:
Diagnostic Test: Endoscopic ultrasound — Upper endoscopy using an echoendoscope to obtain ultrasound images of the pancreaticobiliary system and adjacent structures.

SUMMARY:
We hope to better define the association between opiate use and biliary dilation, which was evident in our previous retrospective study. This prospective study including all endoscopic ultrasound procedures performed for further evaluation of biliary dilatation in the setting of bilirubin <2 mg/dL will enable accurate measurement of common bile duct and pancreatic duct diameter using endoscopic ultrasound and identification of other non- obstructive factors which may modulate biliary dilation (i.e. age, cholecystectomy status, duration and type of opiate used).

DETAILED DESCRIPTION:
We hope to better define the association between opiate use and biliary dilation, which was evident in our previous retrospective study. This prospective study including all endoscopic ultrasound procedures performed for further evaluation of biliary dilatation in the setting of bilirubin <2 mg/dL will enable accurate measurement of common bile duct and pancreatic duct diameter using endoscopic ultrasound and identification of other non- obstructive factors which may modulate biliary dilation (i.e. age, cholecystectomy status, duration and type of opiate used).

We believe this work will be of great interest to gastroenterologists, as it provides additional data for interpretation of isolated common bile duct dilation in asymptomatic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Referral/consultation for consideration for EUS ± ERCP
2. Age 18 and older
3. Evidence of biliary dilation on abdominal imaging without obstructive pattern on liver function tests or imaging.
4. Willing and able to comply with the study procedures and provide written informed consent to participate in the study.

Exclusion Criteria:

1. Age <18
2. Potentially vulnerable subjects including, homeless people, pregnant females, employees and students.
3. Participation in another investigational study that may directly or indirectly affect the results of this study within 30 days prior to the initial visit
4. Other biliary process which accounts for patient's abnormal liver function studies/imaging (i.e. mass, stone, cirrhosis).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred for endoscopic ultrasound (EUS) or endoscopic retrograde cholangiopancreatography (ERCP) for further evaluation of abnormal imaging findings will be screened for inclusion in this study. Patients with biliary dilatation who meet all the inclusion criteria and have none of the exclusion criteria will be invited to participate in this prospective study during their initial clinic visit or hospital consultation.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01-03 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Identification of factors associated with biliary dilation | Up to 3 hours
  Statistical analysis will be conducted to assess for association between opiate use (including type and duration of opiates) and common bile duct diameter. We will also evaluate for other factors predictive of increased common bile duct diameter, which may include age and cholecystectomy status (based on our initial retrospective study). Power calculations to determine sample size were extrapolated from the initial retrospective study at our institution.
Identification of factors associated with pancreatic duct dilation | Up to 3 hours
  Statistical analysis will be conducted to assess for association between opiate use (including type and duration of opiates) and common bile duct diameter. We will also evaluate for other factors predictive of increased common bile duct diameter, which may include age and cholecystectomy status (based on our initial retrospective study). Power calculations to determine sample size were extrapolated from the initial retrospective study at our institution.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University Medical Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No